CLINICAL TRIAL: NCT06216041
Title: A Phase I, Single-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of IMM-H014 Sand the Effects of Food on Pharmacokinetics in Healthy Subjects
Brief Title: To Evaluate the Safety, Tolerability, Pharmacokinetics and Food Effects of IMM-H014 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun Intellicrown Pharmaceutical Co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-I-IMM-H014-01
Record Dates: First submitted 2024-01-03; First posted 2024-01-22 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
Keywords: Adverse Event
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking for Participant, Investigator and Clinical Research Associate
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- IMM-H014 /Placebo(single dose) 12.5 mg (Cohort 1) (Experimental): IMM-H014 /Placebo tablets administered orally once daily under fasted condition.
  Interventions: Drug: IMM-H014; Drug: Placebo
- IMM-H014 /Placebo((single dose) 37.5 mg Cohort(Cohort 2) (Experimental): IMM-H014 /Placebo tablets administered orally once daily under fasted condition.
  Interventions: Drug: IMM-H014; Drug: Placebo
- IMM-H014 /Placebo(single dose) 75 mg (Cohort 3) (Experimental): IMM-H014 /Placebo tablets administered orally once daily under fasted condition.
  Interventions: Drug: IMM-H014; Drug: Placebo
- IMM-H014 /Placebo(single dose) 125 mg(Cohort 4) (Experimental): IMM-H014 /Placebo tablets administered orally once daily under fasted condition.
  Interventions: Drug: IMM-H014; Drug: Placebo
- IMM-H014 /Placebo(single dose and food effect) 175mg (Cohort 5) (Experimental): Period 1 (Day1 to Day4): Group A and Group B receive IMM-H014 /Placebo under the fasting or fed condition ,respectively on Day1.
  Period 2 (Day 8 to Day11): Group A and Group B receive IMM-H014 /Placebo under the fed or fasting condition ,respectively on Day8.
  Interventions: Drug: IMM-H014 ( FE); Drug: Placebo ( FE)
- IMM-H014 /Placebo(single dose) 225 mg (Cohort 6) (Experimental): IMM-H014 /Placebo tablets administered orally once daily under fasted condition.
  Interventions: Drug: IMM-H014; Drug: Placebo
- IMM-H014 /Placebo(single dose) 275mg (Cohort 7) (Experimental): IMM-H014 /Placebo tablets administered orally once daily under fasted condition.
  Interventions: Drug: IMM-H014; Drug: Placebo
- IMM-H014 /Placebo(single dose) 325 mg (Cohort 8) (Experimental): IMM-H014 /Placebo tablets administered orally once daily under fasted condition.
  Interventions: Drug: IMM-H014; Drug: Placebo
- IMM-H014 /Placebo(multiple dose) tentative 37.5 mg(Cohort 9) (Experimental): IMM-H014 /Placebo tablets administered orally once daily under fasted condition for 7 Days(a total of 7 doses).
  Interventions: Drug: IMM-H014; Drug: Placebo
- IMM-H014 /Placebo(multiple dose) tentative 75 mg(Cohort 10) (Experimental): IMM-H014 /Placebo tablets administered orally once daily under fasted condition for 7 Days(a total of 7 doses).
  Interventions: Drug: IMM-H014; Drug: Placebo
- IMM-H014 /Placebo(multiple dose) tentative 125 mg(Cohort 11) (Experimental): IMM-H014 /Placebo tablets administered orally once daily under fasted condition for 7 Days(a total of 7 doses).
  Interventions: Drug: IMM-H014; Drug: Placebo
- IMM-H014 /Placebo(multiple dose) tentative 175 mg(Cohort 12) (Experimental): IMM-H014 /Placebo tablets administered orally once daily under fasted condition for 7 Days(a total of 7 doses).
  Interventions: Drug: IMM-H014; Drug: Placebo
- IMM-H014 /Placebo(multiple dose) tentative 225 mg(Cohort13) (Experimental): IMM-H014 /Placebo tablets administered orally once daily under fasted condition for 7 Days(a total of 7 doses).
  Interventions: Drug: IMM-H014; Drug: Placebo

INTERVENTIONS:
Drug: IMM-H014 — SAD and MAD adopt "sentinel method "which 2 healthy subjects first will receive IMM-H014, and if are evaluated to be tolerable, the remaining 8 subjects will be randomly assigned to receive IMM-H014 and placebo in a ratio of 3:1(10 in per experimental Cohort).
  Arms: IMM-H014 /Placebo((single dose) 37.5 mg Cohort(Cohort 2); IMM-H014 /Placebo(multiple dose) tentative 125 mg(Cohort 11); IMM-H014 /Placebo(multiple dose) tentative 175 mg(Cohort 12); IMM-H014 /Placebo(multiple dose) tentative 225 mg(Cohort13); IMM-H014 /Placebo(multiple dose) tentative 37.5 mg(Cohort 9); IMM-H014 /Placebo(multiple dose) tentative 75 mg(Cohort 10); IMM-H014 /Placebo(single dose) 12.5 mg (Cohort 1); IMM-H014 /Placebo(single dose) 125 mg(Cohort 4); IMM-H014 /Placebo(single dose) 225 mg (Cohort 6); IMM-H014 /Placebo(single dose) 275mg (Cohort 7); IMM-H014 /Placebo(single dose) 325 mg (Cohort 8); IMM-H014 /Placebo(single dose) 75 mg (Cohort 3)
Drug: Placebo — SAD and MAD adopt "sentinel method "which 2 healthy subjects first will receive IMM-H014, and if are evaluated to be tolerable, the remaining 8 subjects will be randomly assigned to receive IMM-H014 and placebo in a ratio of 3:1(10 in per experimental Cohort).
  Arms: IMM-H014 /Placebo((single dose) 37.5 mg Cohort(Cohort 2); IMM-H014 /Placebo(multiple dose) tentative 125 mg(Cohort 11); IMM-H014 /Placebo(multiple dose) tentative 175 mg(Cohort 12); IMM-H014 /Placebo(multiple dose) tentative 225 mg(Cohort13); IMM-H014 /Placebo(multiple dose) tentative 37.5 mg(Cohort 9); IMM-H014 /Placebo(multiple dose) tentative 75 mg(Cohort 10); IMM-H014 /Placebo(single dose) 12.5 mg (Cohort 1); IMM-H014 /Placebo(single dose) 125 mg(Cohort 4); IMM-H014 /Placebo(single dose) 225 mg (Cohort 6); IMM-H014 /Placebo(single dose) 275mg (Cohort 7); IMM-H014 /Placebo(single dose) 325 mg (Cohort 8); IMM-H014 /Placebo(single dose) 75 mg (Cohort 3)
Drug: IMM-H014 ( FE) — FE part is divided into two groups: 8 subjects will receive IMM-H014 and 2 subjects will receive placebo In group A .All 8 subjects will receive IMM-H014 in group B. Group A adopts "sentinel method ".The treatment in food effect consists of 2 periods.
  Arms: IMM-H014 /Placebo(single dose and food effect) 175mg (Cohort 5)
Drug: Placebo ( FE) — FE part is divided into two groups: 8 subjects will receive IMM-H014 and 2 subjects will receive placebo In group A .All 8 subjects will receive IMM-H014 in group B. Group A adopts "sentinel method ".The treatment in food effect consists of 2 periods.
  Arms: IMM-H014 /Placebo(single dose and food effect) 175mg (Cohort 5)

SUMMARY:
This study will evaluate the safety, tolerability and pharmacokinetics (PK) of escalating single- and multiple-oral doses of IMM-H014 on fasted condition, and characterize PK of IMM-H014 on an empty stomach (fasted condition) and following a high fat, high calorie meal (fed condition) in a 2-period, 2-sequence manner. The study will be conducted in 3 parts (Ascending single dose, multiple dose and food effect). Participants will receive either IMM-H014 or placebo.

DETAILED DESCRIPTION:
The study is a randomized, double-blind phase 1 trial including 3 parts: single ascending dose (SAD) part, multiple ascending dose (MAD) part and food effect (FE) part.

SAD and MAD parts adopt "sentinel method "which2 healthy subjects first will receive IMM-H014, and if are evaluated to be tolerable, the remaining 8 subjects will be randomly assigned to receive IMM-H014 and placebo in a ratio of 3:1(10 in per experimental Cohort). Subjects in SAD will receive 12.5,37.5,75, 125, 225, 275, 325mg (Cohort 1-4 and Cohort 6-8) once daily respectively. Subjects in MAD will receive 37.5, 75, 125, 175, 225mg (Cohort 9 - Cohort 13) once daily for 7days respectively.

FE part is divided into two groups: 8 subjects will receive IMM-H014 and 2 subjects will receive placebo In group A .All 8 subjects will receive IMM-H014 in group B. Group A adopts "sentinel method ".The treatment in food effect consists of 2 periods, and subjects will receive175mg(SAD Cohort 5) on fasting and postprandial states respectively. There will be a 7-day wash out period between treatment periods. To monitor AEs, record abnormalities (12-lead ECG, Vital signs, Physical examination, Clinical Laboratory), and detect the pharmacokinetics of IMM-H014.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects can voluntarily participate in the clinical trial, sign informed consent before the trial, fully understand the trial content, process and possible adverse events, and complete the study in accordance with the requirements of the trial protocol;
2. Subjects can use effective contraceptive methods, such as abstinence, condoms, IUD use, and dual barrier method (such as condom plus diaphragm), within 6 months from the beginning of screening to the last trial drug administration;
3. 18-45 years of age, male and female (including 18 and 45 years);
4. Male weight ≥50kg, female weight ≥45kg; Body mass index (BMI) in the range of 18-28 kg/m2 (including the cut-off value); 5）Vital signs and physical examination with normal or abnormal has no clinical significance.

Exclusion Criteria:

1. Clinical history of drug allergy or specific allergic diseases (asthma, urticaria), or known or suspected allergic history to experimental drugs and related excipients;
2. Subjects who have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines and health products within 2 weeks before screening;
3. Clinical laboratory examination (blood routine, urine routine, blood biochemistry, coagulation function, virology examination, thyroid function), abdominal color Doppler ultrasound (liver, gallbladder, spleen, pancreas, kidneys, adrenal gland), chest radiography and other abnormalities with clinical significance; Or other clinically significant diseases (including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular diseases) within 6 months before screening;
4. Subjects who ate diets (including grapefruit or grapefruit products, pitaya, mango, etc.) that may affect drug metabolism within 7 days before screening, or had strenuous exercise, or the researchers thought that there were other dieters that affected drug metabolism, absorption, distribution, metabolism and excretion;
5. A family history of a first-degree relative (i.e., biological parent, sibling, or child) with a risk factor for tip torsional ventricular tachycardia, or a family history of short QT syndrome, long QT syndrome, sudden unexplained death in youth (less than/etc. 40 years old), or sudden infant death syndrome;
6. Subjects who suffer from hyperkalemia, hypokalemia, hypermagnesemia, hypomagnesemia, hypercalcemia or hypocalcemia which are abnormal and clinically significant by the investigator;
7. Presence of clinically significant abnormalities in ECG or QTcF>450ms (corrected according to Frederica formula, the calculation method is QTCF = Qt/(RR 0.33));
8. Creatinine clearance rate < 90mL/min (Creatinine clearance calculation Cockcroft-Gault formula: CrCl = [(140 - age) by weight (kg)] / [0.814 x Scr (umol/L)] or CrCl = (140 - age) by weight (kg) / 72 x Scr (mg/dL), women need to according to the formula calculation results by 0.85);
9. Suffering from chronic or active gastrointestinal diseases, such as esophageal diseases, acute gastritis, gastric and duodenal ulcers, enteritis, active gastrointestinal bleeding, or gastrointestinal surgery, which investigators believe is still clinically relevant;
10. Subjects who had undergone major surgery (excluding diagnostic surgery) in the six months prior to screening, or who will undergo surgery during the study period, or who had undergone surgery that the investigator determines will affect drug absorption, distribution, metabolism, or excretion;
11. Participants who had participated in other clinical trials within 3 months prior to screening (participants can be enrolled if they withdraw from the study before administration of the investigational drug, that is, they have not received the drug);
12. Blood donation or significant blood loss (> 450ml) within 3 months prior to screening;
13. Had a history of alcohol abuse (drinking an average of 14 units of alcohol per week in the 3 months prior to screening (1 unit =360 mL beer or 45mL liquor with 40% alcohol or 150 ml wine), or could not abstinence during the test period, or had a positive alcohol breath test;
14. Smoking more than 5 cigarettes per day in the 3 months before screening;
15. Have a history of drug or drug abuse or urine drug abuse screening positive;
16. Subjects who have special requirements for diet and cannot accept a unified diet;
17. Have dysphagia;
18. Female subjects are lactating or have positive serological pregnancy results.
19. Acute illness or concomitant medication occurred between the screening stage and the administration of the investigational drug;
20. Ingested chocolate, any food or drink containing caffeine or rich in xanthines within 24 hours before first taking the experimental drug;
21. Subjects who taken any alcohol-containing product or a positive alcohol breath test in the 24 hours prior to the use of the study drug;
22. The investigator believes that the subjects are not suitable to participate in the clinical study for other reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events following oral doses (single, multiple and food effect)of IMM-H014 and placebo | through study completion, up to 11, 17, 18 days for SAD, MAD, FE part
  the adverse events are recorded according to the actual occurrence
Number of participants with abnormal laboratory tests results and abnormal physical exam findings | through study completion, up to 4, 10, 11 days for SAD, MAD, FE part
  The data of the clinical research center is collected and analyzed according to the time point of the test flow chart

SECONDARY OUTCOMES:
PK parameters: AUClast（AUC0-t） | Up to 4, 10, 11 days for SAD, MAD, FE part
  AUClast is defined as the concentration of drug from time zero to the last quantifiable concentration.
PK parameters: AUCinf（AUC0-∞） | Up to 4, 10, 11 days for SAD, MAD, FE part
  AUCinf is defined as the concentration of drug extrapolated to infinite time (area under the plasma concentration versus time curve extrapolated to infinite time).
PK parameters: Cmax | Up to 4, 10, 11 days for SAD, MAD, FE part
  Cmax is defined as the maximum observed concentration of drug in plasma.
PK parameters: Tmax | Up to 4, 10, 11 days for SAD, MAD, FE part
  Tmax is defined as the time to maximum concentration.
PK parameters: t1/2 | Up to 4, 10, 11 days for SAD, MAD, FE part
  t1/2z is defined as the time to decline half of the drug concentration in plasma.
PK parameters: CL/F | Up to 4, 10, 11 days for SAD, MAD, FE part
  λz is defined as the ratio between the elimination of compound per unit time and the total amount of compound.
PK parameters: λz | Up to 4, 10, 11 days for SAD, MAD, FE part
  λz is defined as the ratio between the elimination of compound per unit time and the total amount of compound.
Multiple-dose plasma PK parameter: Rac | Up to 10 days
  Rac (Accumulation Index) is defined as the ratio between AUC0-XX in Day XX and AUC0-XX in Day1
Multiple-dose plasma PK parameter: DF | Up to 10 days
  DF is defined as the percentage of fluctuation in steady state is 100 * (Cmax, ss - Cmin, ss)/Cavg, ss
Multiple-dose plasma PK parameter: Cmin | Up to 10 days
  Cmin is defined as the minimum observed concentration of drug in plasma at steady state.
Multiple-dose plasma PK parameter: Cmax | Up to 10 days
  Cmax is defined as the maximum observed concentration of drug in plasma at steady state.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The first Bethune hospital of Jilin University, Changchun, Jilin, China